CLINICAL TRIAL: NCT01356056
Title: Tele-diagnostics for Remote Parkinson's Monitoring
Status: Completed | Type: Observational
Sponsor: Great Lakes NeuroTechnologies Inc. (Industry)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 10-09-29-03EE; 7R43NS065554-03 (NIH); 5R43MD004049-02 (NIH)
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Kinesia HomeView Monitoring: Uses Kinesia HomeView at home once per week
  Interventions: Device: Kinesia HomeView
- Control: Assessed in the clinic every 4 weeks using traditional methods

INTERVENTIONS:
Device: Kinesia HomeView — Quantifies motor symptom severity in the home
  Groups: Kinesia HomeView Monitoring

SUMMARY:
The purpose of this research study is to design, implement, and clinically assess a portable, user worn system for monitoring Parkinson's disease (PD) motor symptoms. The current standard in evaluating symptoms is the Unified Parkinson's Disease Rating Scale (UPDRS), a subjective, qualitative ranking system. The main goal of this research is to develop a quantitative system, Kinesia HomeView, to assess tremor as well as different features of bradykinesia in a home based system which can capture those symptom changes over the course of a day and aid in evaluating treatment protocol efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Parkinson's disease

Exclusion Criteria:

* Inability to follow the required clinical instruction
* Subjects with cognitive impairments that would prohibit them from properly using the Kinesia HomeView system
* Subjects without the cognitive ability to respond to researchers and let them know when any parameters of the study may become uncomfortable
* Subjects found on examination by our clinicians to have any physical limitations which would be counter productive to participation in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
UPDRS | Every 4 weeks
PDQ-39 | Every 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States